CLINICAL TRIAL: NCT02829892
Title: Using Environmental Light Therapy to Improve Sleep and Neuropsychiatric Symptoms in Dementia
Acronym: SOLEIL SOMMEIL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 14-PP-16
Record Dates: First submitted 2016-07-08; First posted 2016-07-12 (Estimated); Last update posted 2016-07-12 (Estimated); Status verified 2016-07

CONDITIONS: Polypathology and Autonomy Loss
MeSH Terms: interventions — Phototherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Light therapy (Other): Innovative ambient lighting
  Interventions: Device: Light therapy

INTERVENTIONS:
Device: Light therapy — 14-days exposure with an innovative ambient light

SUMMARY:
Alzheimer's disease and related syndromes (AD) is a disease affecting memory but also the relationship with the environment and empower people. Patients with AD present in 90% of cases of behavioral disorders and of these behavioral disorders include agitation, apathy but also sleep disorders by circadian rhythm impairment.. No study has shown proven efficacy on the behavior of patients with AD. The main objective of the study was to assess the influence of environmental light nighttime sleep of residents.

DETAILED DESCRIPTION:
Alzheimer's disease and related syndromes (AD) is a disease affecting memory but also the relationship with the environment and empower people. Patients with AD present in 90% of cases of behavioral disorders and of these behavioral disorders include agitation, apathy but also sleep disorders by circadian rhythm impairment. In 2014, the Cochrane published a systematic review of the literature over the last 20 years concerning the use of light therapy in patients with a AD. No study has shown proven efficacy on the behavior of patients with AD. The main objective of the study was to assess the influence of environmental light therapy (from 5 a.m to 10 p.m) on nighttime sleep of residents. Secondary objectives were the study of sleep time on the day, anxiety by the COVI scale and behavioral disorders by the NPI scale.

ELIGIBILITY:
Inclusion Criteria:

* EHPAD residents at Les Pastoureaux Valenton having moderate to severe MASA
* More than 60 years
* Presenting motor behavioral disorders and / or anxiety and / or restlessness and / or insomnia .
* No underlying acute medical problems including no delirium

Exclusion Criteria:

* Residents refusing to lend to experimentation
* Resident who are not matching with the inclusion criteria
* total acquired or congenital blindness
* bedridden patient ( loss of physical autonomy)
* Entry to the residence less than 15 days before the start of the experiment.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2015-06; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Sleep duration between 10 p.m to 5 a.m | 14 days

SECONDARY OUTCOMES:
Sleep duration by day | 14 days
Number of awake between 10 p.m to 5 a.m | 14 days
Anxiety by the COVI scale | 14 days
Behavioral disorders by the NPI scale | 14 days

CONTACTS AND LOCATIONS:
Locations (1):
- EHPAD ORPEA Valenton, Valenton, France

IPD SHARING:
Plan to Share IPD: Undecided